CLINICAL TRIAL: NCT02746055
Title: Cross-Sectional Study of the Prevalence of TGFBI Corneal Dystrophies
Brief Title: Study of the Prevalence of TGFBI Corneal Dystrophies
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Avellino Labs USA, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Avel2016PS
Record Dates: First submitted 2016-04-15; First posted 2016-04-21 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Corneal Dystrophy
MeSH Terms: conditions — Corneal Dystrophies, Hereditary

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — buccal epithelial swabs
Oversight: Data Monitoring Committee: No

SUMMARY:
To determine the prevalence of 5 specific corneal dystrophies in a subgroup of patients seeking refractive surgery, and to use that information to inform them and their refractive surgeons of the presence of the corneal dystrophies so that they may make safer choices when considering refractive surgery.

DETAILED DESCRIPTION:
It is well established in the peer-reviewed literature that elective keratorefractive surgery is contraindicated in individuals with granular corneal dystrophy type 2 (GCD2).1,2,3,4 Although all reported cases of exacerbation of dystrophic stromal deposits have been in individuals with GCD2, it may be assumed that a similar accelerated deposition would occur in individuals with any of the TGFBI dystrophies, and thus elective keratorefractive surgery should be avoided in any individual with a TGFBI dystrophy. The commercially available Avellino Refractive Surgery Safety Test (Avellino Universal Test) offers an accurate, rapid and affordable way to screen for five corneal dystrophies associated with mutations in the TGFBI gene prior to keratorefractive surgery. These dystrophies are granular dystrophy type 1 (GCD1), GCD2, lattice corneal dystrophy type 1 (LCD1), Reis-Buckler corneal dystrophy, and Thiel- Behnke corneal dystrophy.

This is a multicenter, cross-sectional, observational study of the prevalence of TGFBI corneal dystrophies in a North American population. Patients presenting to the clinical site for an ocular examination with a refractive complaint (non-medical complaint) or for refractive surgery consultation will be asked to participate in this study. Prior to the collection of any study data, Informed Consent will be obtained.

A a serial number / bar code controlled case report form (CRF) single nucleotide variants implicated in the pathogenesis of the TGFBI corneal dystrophies. The CRF will be used to collect demographic information from the patient. Slit lamp examination of the corneas will be performed, and the presence or absence of corneal opacities, whether characteristic or not of a TGFBI dystrophy, will be documented on the CRF form.

Once all data has been collected, descriptive statistics will be computed to identify the prevalence of each of the TGFBI corneal dystrophies as defined by the genotype. Demographic data will be compared between unaffected individuals and those identified to have a coding region mutation associated with one of the five aforementioned TGFBI corneal dystrophies.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Able and willing to provide written informed consent and sign a HIPAA form.

Exclusion Criteria:

• None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the clinical site for refractive surgery consultation or routine ocular examination who are:
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-12 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Prevalence of the genetic mutations in the TGFBI gene will be measured by using buccal epithelium and real time PCR-based genetic analysis. | One year
  Descriptive statistics will be computed to identify prevalence of each of the TGFBI corneal dystrophies as defined by the genotype. Demographic data will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony J Aldave, MD, Study Director — UCLA Stein Eye Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aldave AJ, Sonmez B, Forstot SL, Rayner SA, Yellore VS, Glasgow BJ. A clinical and histopathologic examination of accelerated TGFBIp deposition after LASIK in combined granular-lattice corneal dystrophy. Am J Ophthalmol. 2007 Mar;143(3):416-9. doi: 10.1016/j.ajo.2006.11.056. Epub 2006 Dec 29. PMID 17317389
- [Background] Banning CS, Kim WC, Randleman JB, Kim EK, Stulting RD. Exacerbation of Avellino corneal dystrophy after LASIK in North America. Cornea. 2006 May;25(4):482-4. doi: 10.1097/01.ico.0000195949.93695.37. PMID 16670492
- [Background] Roh MI, Grossniklaus HE, Chung SH, Kang SJ, Kim WC, Kim EK. Avellino corneal dystrophy exacerbated after LASIK: scanning electron microscopic findings. Cornea. 2006 Apr;25(3):306-11. doi: 10.1097/01.ico.0000183536.07275.9a. PMID 16633031
- [Background] Jun RM, Tchah H, Kim TI, Stulting RD, Jung SE, Seo KY, Lee DH, Kim EK. Avellino corneal dystrophy after LASIK. Ophthalmology. 2004 Mar;111(3):463-8. doi: 10.1016/j.ophtha.2003.06.026. PMID 15019320
- [Background] Lee JH, Cristol SM, Kim WC, Chung ES, Tchah H, Kim MS, Nam CM, Cho HS, Kim EK. Prevalence of granular corneal dystrophy type 2 (Avellino corneal dystrophy) in the Korean population. Ophthalmic Epidemiol. 2010 Jun;17(3):160-5. doi: 10.3109/09286581003624939. PMID 20455845
- [Background] Lakshminarayanan R, Chaurasia SS, Anandalakshmi V, Chai SM, Murugan E, Vithana EN, Beuerman RW, Mehta JS. Clinical and genetic aspects of the TGFBI-associated corneal dystrophies. Ocul Surf. 2014 Oct;12(4):234-51. doi: 10.1016/j.jtos.2013.12.002. Epub 2014 Jul 18. PMID 25284770